CLINICAL TRIAL: NCT01798823
Title: Exercise-induced Bronchoconstriction in School Children - Prevalence, Environmental/Individual Risk Factors and Its Mechanism
Brief Title: Exercise-induced Bronchoconstriction in School Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Iwona Stelmach, MD, PhD, Prof., Medical University of Lodz
Other Study IDs: RNN/160/12/KE
Record Dates: First submitted 2013-02-19; First posted 2013-02-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Asthma
Keywords: children; asthma
MeSH Terms: conditions — Asthma | interventions — Health Records, Personal; Restraint, Physical; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * exhaled breath condensate sample
  * blood sample (5 ml sample): tryptase, lipoxin A4 serum levels
  * blood sample also will be taken before and after challenge together with exhaled breath condensate sample in order to detect markers of inflammation (such as IL-1a, IL-2, IL-5, IL-6, IL-8, IL-9, IL-12p70, IL-13, IL-17, IL-22, MCP1, TLR2, MIP1a, PDGFBB, TIMP2, TNFalfa, CRP, TGF-b1, TSLP- ELISA and cysteinyl leukotrienes, LTB4, PGE2-HPLC/mass spectrometry).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- EIB+A+: * children with EIB and asthma
  * History, physical, LF, SPT, blood sample, FeNO, EBC
  Interventions: Procedure: History, physical, LF, SPT, blood sample, FeNO, EBC.
- EIB+A-: * children with EIB without asthma
  * History, physical, LF, SPT, blood sample, FeNO, EBC
  Interventions: Procedure: History, physical, LF, SPT, blood sample, FeNO, EBC.
- EIB-A+: * children without EIB and asthma
  * History, physical, LF, SPT, blood sample, FeNO, EBC
  Interventions: Procedure: History, physical, LF, SPT, blood sample, FeNO, EBC.
- EIB-A-: * children without EIB without asthma
  * History, physical, LF, SPT, blood sample, FeNO, EBC
  Interventions: Procedure: History, physical, LF, SPT, blood sample, FeNO, EBC.

INTERVENTIONS:
Procedure: History, physical, LF, SPT, blood sample, FeNO, EBC. — Medical history and physical examination, (LF) lung function (spirometry, (SETC) standardized exercise treadmill challenge, (BRT) bronchial reversibility test,(MBP) metacholine bronchial provocation), (SPT) skin prick tests, blood sample, (FeNO) fractional exhaled nitric oxide measurements, (EBC) exhaled breath condensate.

SUMMARY:
The goal of the project is to define the prevalence and inflammatory background of exercise-induced bronchoconstriction (EIB) in school children and determine individual and environmental risk factors for EIB. The obtained results will provide objective measures on biological processes leading to bronchoconstriction during exercise, as might be experienced naturally during the school life. The results could be applied in the management of EIB patients with or without asthma. The results of planned research will be published in journals with national and international impact, and presented during symposia and conferences.

DETAILED DESCRIPTION:
Methods:

Patients and Study design It will be two-step study carried out among school teenagers. In the first step the school children will be screened for EIB during physical education (PE) lesson. Inn all children before and after physical exercise (PE) lesson spirometry will be performed. Children with decreased FEV1 (>=10% from baseline) and/or children with EIB history within last 12 months (symptoms: dyspnea, cough, wheezes, chest pain during/after exercises) will be invited to the clinic for future evaluation and qualified to the next step of the study.

In the second step children with suspected EIB and their parents will be invited to the clinic. Three visits are planned. Treatment with long acting beta agonists will be stopped 24 hours before each visit; antihistamine treatment will be stopped 21 days before the first visit.

First visit

In all children standardized exercise trade mil challenge together with reversibility test and skin prick tests will be performed. Based on these results children will be divided to the following groups:

* children with EIB and asthma (EIB+A+)
* children with EIB without asthma (EIB+A-)
* children without EIB and asthma (EIB-A+)
* children without EIB without asthma (EIB-A-) Second visit Twenty children will be randomly selected from each group. In all children standardized exercise trade mil challenge will be performed again together. Blood sample will be taken before and after challenge together with exhaled breath condensate sample in order to detect markers of inflammation. Also before and after exercise challenge exhaled nitric oxide will be measured.

Third visit Bronchial provocation challenge with metacholine will be performed in each child.

Methods

* medical history and physical examination
* lung function tests Pulmonary function tests Pulmonary function testing will be performed with a Master Screen unit (Erich Jaeger Gmbh-Hochberg, Germany). Predicted values for all lung function variables are based on a previous study of healthy controls provided by the manufacturer of the lung function test equipment. Flow-volume curves will be performed according to the American Thoracic Society standards. The highest of 3 successful measurements will be taken and analyzed. The results will be expressed as the percentage of a predicted value. All the subjects will be able to perform spirometry.
* exhaled nitric oxide measurements The NO measurements will be performed according to European Respiratory Society/American Thoracic Society (ERS/ATS) recommendations with a chemiluminescence analyzer (model 280i nitric oxide analyzer; Sievers, Boulder, CO, USA) and deaned in parts per billion. The analyzer provides an on-line continuous measurement of NO in a single exhalation with a detection range of 0.1 to 500 ppb. Environmental NO will be measured before and after each test and never exceed 5 ppb. All subjects are studied in the sitting position, without wearing a nose clip. The subjects exhale at a constant ﬂow rate (50mL/s) from total lung capacity to residual volume without breath holding. They maintain a constant mouth pressure (17 cm H2O) by monitoring a visual display in order to eliminate contamination from nasal NO. Dead space and nasal NO (which are reﬂected by the NO concentration peak during exhalation) and NO from the lower respiratory tract (determined by the plateau value after the peak) are recorded automatically by using the manufacturer's software. Three fractional exhaled nitric oxide (FeNO) measurements of the plateau phase will be obtained, with less than 10% variation. The mean value of 3 successive, reproducible recordings will be retained for statistical analysis.
* standardized exercise treadmill challenge Exercise-induced bronchoconstriction will be tested by the use of a motor-driven treadmill (Kettler, Ense-Parsit, Germany) according to ATS/ERS guidelines. The children will be instructed to run for 8 minutes with a submaximal exercise load. The exercise test consist of a 2-minute warm-up and 6 minutes of steady-state running on a treadmill inclined to produce a heart rate of at least 95% of the maximum predicted for age (calculated as 220 - age [years]). The slope of the treadmill is 5.5% (3°). Small adjustments in workload (treadmill speed) will be made, if necessary, to achieve targeted hearth rates. Nasal clips will be used during the test, and heart rate will be continuously monitored (electronic heart rate scanner; Kettler). The submaximal run on the treadmill will be performed at the same speed (exercise load) on both test occasions (at randomization and after 4 weeks of treatment) for each child. The ambient temperature in the air-conditioned laboratory will be kept stable at 22°C, and the humidity will be stable between 40% and 50% on each day of the study. Differences of 1°C in temperature and 5 mg H2 OxL-1 of air humidity on the test days on each patient will be accepted. 14 FEV1 will be measured before running, immediately after, and 3, 6, 10, 15, 20 and 30 minutes after running. Maximum percentage fall in FEV1 after exercise test will be calculated by using the following formula: [(pre-exercise FEV1 - lowest postexercise FEV1) /pre-exercise FEV1] x 100. The FEV1 values will be plotted against time for each treatment. The area under the curve (AUC) for the FEV1 values from exercise over the 30-minute period will be calculated by using a trapezoidal rule. EIB will be defined as a ≥ 15% decrease in FEV1 from baseline within the first 5 minutes after exercise.
* exhaled breath condensate EBC samples will be collected through EcoScreen-II device (Viasys Healthcare GmbH, Berlin, Germany). Samples of exhaled breath condensate (EBC) will be obtained from children during tidal breathing while wearing a nose clip, as describe previously [6]. The two-way non-rebreathing valves and tubing to the condenser will be served as a saliva trap. After collection (during 10min), EBC will be rapidly frozen in small plastic tubes at -80°C using dry ice and will be stored at -80°C until analysis.

The material will be the exhaled breath condensate of children diagnosed with asthma. The analysis will be performed using Quantibody Human Inflammation Array 3 (RayBiotech, Norcross, GA, USA) according to the manufacturer's instructions. This multiplex ELISA array kit allows quantitative measurement of 40 human cytokines. Each standard glass slide consists of 16 wells, each with an identical cytokine antibody array. All antibodies and positive controls will be printed in quadruplicated in every well.

In the first step, the capture antibody is bound to the glass surface of the slide. Next, 100 µl of each patient sample and the aray specific cytokine standards of known concentration are added to each well. After incubation for 2 hours at the room temperature, the array is washed 5 times with 150 µl of Wash Buffer I and twice with 150 µl of Wash Buffer II, 5 minutes per wash. Next, the array is incubated for 2 hours with 1.4 ml of the biotin - conjugated antibody at the room temperature. Then the washing protocol is repeated before the addition of 80 µl of Cy3 equivalent dye-conjugated streptavidin to each well for 1 hour. After washing the array, the fluorescence signal is detected and quantified with the Axon GenePix 4000B scanner and GenePix Pro 6.0 software (Molecular Devices). The results will be analyzed using Q - Analyzer Software (RayBiotech, Norcross, GA, USA).

* metacholine bronchial provocation challenge Metacholine bronchial test of the provocation will be performed using the dosimeter technique aerosol provocation system (APS) Pro (Erich Jaeger Gmbh-Hochberg, Germany) with controlled tidal breathing. After the pulverization physiological diluent, methacholine will be delivered in four cumulative doses: 0,015 mg, 0,045mg, 0,18mg, 0,72mg. Metacholine based provocation test (MBPT) is continued with 2-min intervals between the inhalations until a fall in forced expiratory volume in 1s (FEV1) of ≥20% will be obtained. Provocative dose (PD20) is calculated by linear interpolation on a log-dose-response curve (13).
* in blood sample (5 ml sample): tryptase, lipoxin A4 serum levels
* also in the present study blood sample will be taken before and after challenge together with exhaled breath condensate sample in order to detect markers of inflammation (such as interleukin (IL)-1a, IL-2, IL-5, IL-6, IL-8, IL-9, IL-12p70, IL-13, IL-17, IL-22, monocyte chemoattractant protein one (MCP1), toll-like receptor 2 (TLR2),macrophage inflammatory protein one alfa (MIP1a), platelet derived growth factor (PDGFBB), tissue inhibitor of metalloproteinase two (TIMP2), tumor necrosis factor alpha (TNFalpha), C reactive protein (CRP), transforming growth factor beta one (TGF-b1), thymic stromal lymphopoietin (TSLP) - ELISA and cysteinyl leukotrienes, leukotriene B4 (LTB4), prostaglandin E2 - high pressure liquid chromatography ((PGE2-HPLC))/mass spectrometry).

Meaning:

Practical assessment/The results of proposed study will allow us to assess the prevalence and define the inflammatory background of exercise-induced bronchoconstriction (EIB) in school children. School absence, morbidity, and co-morbidity affecting physical activity will be verified and undiagnosed patients will be treated. Significance of environmental (tobacco smoking, type of exercise, temperature and humidity of exercise room) and individual (age, gender, atopy, obesity, recurrent respiratory truck infections, presence of chronic diseases) factors will be verified.

New findings/Main findings of study will allow to define primary prevention methods of EIB without exercise avoidance, and new recommendations for EIB treatment in children:

1. EIB screening in real live environment (during exercise lesson at school) verified by standardized exercise test in the clinic
2. Defining the individual and environmental risk factors of EIB in school children
3. Kinetics of inflammatory markers (in exhaled breath condensate and serum) during exercise test
4. Complex evaluation of clinical and inflammatory profile of patients with EIB with/without asthma.

Findings in the field/To define markers of inflammation in EIB and possible differences between asthmatic and non-asthmatic children with/without EIB.

Effects/The goal of the project is to define the prevalence and inflammatory background of exercise-induced bronchoconstriction (EIB) in school children and determine individual and environmental risk factors for EIB. The obtained results will provide objective measures on biological processes leading to bronchoconstriction during exercise, as might be experienced naturally during the school life. The results could be applied in the management of EIB patients with or without asthma. The results of planned research will be published in journals with national and international impact, and presented during symposia and conferences.

ELIGIBILITY:
Inclusion Criteria:

* Children with decreased FEV1 (>=10% from baseline) and/or children with EIB history within last 12 months (symptoms: dyspnea, cough, wheezes, chest pain during/after exercises)

Exclusion Criteria:

* Children without decreased FEV1 (>=10% from baseline) and/or children without EIB history within last 12 months (symptoms: dyspnea, cough, wheezes, chest pain during/after exercises)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: school-children screened for EIB during PE lesson
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
- Prevalence and inflammatory background of exercise-induced bronchoconstriction (EIB) in school children, individual and environmental risk factors for EIB | 26 days (maximal)
  - prevalence and inflammatory background of exercise-induced bronchoconstriction (EIB) in school children, individual and environmental risk factors for EIB: Medical history and physical examination, (LF) lung function (spirometry, (SETC) standardized exercise treadmill challenge, (BRT) bronchial reversibility test,(MBP) metacholine bronchial provocation), (SPT) skin prick tests, blood sample, (FeNO) fractional exhaled nitric oxide measurements, (EBC) exhaled breath condensate.

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Stelmach, MDPhDProf., Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, N. Copernicus Hospital, Lodz, Poland , 93-513
Locations (1):
- Department of Pediatrics and Allergy, Medical University of Lodz, N. Copernicus Hospital, Lodz, Poland

REFERENCES:
- [Derived] Stelmach I, Sztafiska A, Jerzyska J, Podlecka D, Majak P, Stelmach W. New insights into treatment of children with exercise-induced asthma symptoms. Allergy Asthma Proc. 2016 Nov;37(6):466-474. doi: 10.2500/aap.2016.37.3993. PMID 27931302
- [Derived] Stelmach I, Cichalewski L, Majak P, Smejda K, Podlecka D, Jerzynska J, Stelmach W. School environmental factors are predictive for exercise-induced symptoms in children. Respir Med. 2016 Mar;112:25-30. doi: 10.1016/j.rmed.2016.01.010. Epub 2016 Jan 21. PMID 26847408
- [Derived] Zaczeniuk M, Woicka-Kolejwa K, Stelmach W, Podlecka D, Jerzynska J, Stelmach I. Methacholine challenge testing is superior to the exercise challenge for detecting asthma in children. Ann Allergy Asthma Immunol. 2015 Dec;115(6):481-4. doi: 10.1016/j.anai.2015.09.022. Epub 2015 Oct 23. PMID 26602490
- [Derived] Majak P, Cichalewski L, Ozarek-Hanc A, Stelmach W, Jerzynska J, Stelmach I. Airway response to exercise measured by area under the expiratory flow-volume curve in children with asthma. Ann Allergy Asthma Immunol. 2013 Dec;111(6):512-5. doi: 10.1016/j.anai.2013.08.026. Epub 2013 Sep 25. PMID 24267361